CLINICAL TRIAL: NCT07169240
Title: Evaluation of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BT-114143 Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ScinnoHub Pharmaceutical Co., Ltd. (Industry)
Collaborators: Peking University Care Luzhong Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT-114143-I-001
Record Dates: First submitted 2025-08-17; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Healthy Subjects (HS)
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Dose level S-2 (Experimental)
  Interventions: Drug: BT-114143
- Dose level S-1 (Experimental)
  Interventions: Drug: BT-114143
- Dose level S1 (Experimental)
  Interventions: Drug: BT-114143
- Dose level S2 (Experimental)
  Interventions: Drug: BT-114143
- Dose level S3 (Experimental)
  Interventions: Drug: BT-114143
- Dose level S4 (Experimental)
  Interventions: Drug: BT-114143
- Dose level S5 (Experimental)
  Interventions: Drug: BT-114143
- Dose level S6 (Experimental)
  Interventions: Drug: BT-114143
- Dose level S7 (Experimental)
  Interventions: Drug: BT-114143
- Dose level S8 (Experimental)
  Interventions: Drug: BT-114143
- Dose level S9 (Experimental)
  Interventions: Drug: BT-114143
- control group (Placebo Comparator)
  Interventions: Drug: 0.9% Sodium Chloride Injection as Placebo

INTERVENTIONS:
Drug: BT-114143 — 6 subjects will receive a single dose of BT-114143 injection at 0.03 mg/kg.
  Arms: Dose level S-1
Drug: BT-114143 — 6 subjects will receive a single dose of BT-114143 injection at 0.07 mg/kg.
  Arms: Dose level S-2
Drug: BT-114143 — 3 subjects will receive a single dose of BT-114143 injection at 0.15 mg/kg.
  Arms: Dose level S1
Drug: BT-114143 — 6 subjects will receive a single dose of BT-114143 injection at 0.3 mg/kg.
  Arms: Dose level S2
Drug: BT-114143 — 6 subjects will receive a single dose of BT-114143 injection at 0.6 mg/kg.
  Arms: Dose level S3
Drug: BT-114143 — 6 subjects will receive a single dose of BT-114143 injection at 1.2 mg/kg.
  Arms: Dose level S4
Drug: BT-114143 — 6 subjects will receive a single dose of BT-114143 injection at 2.4 mg/kg.
  Arms: Dose level S5
Drug: BT-114143 — 6 subjects will receive a single dose of BT-114143 injection at 4.8 mg/kg.
  Arms: Dose level S6
Drug: BT-114143 — 6 subjects will receive a single dose of BT-114143 injection at 8.4 mg/kg.
  Arms: Dose level S7
Drug: BT-114143 — 6 subjects will receive a single dose of BT-114143 injection at 12.6 mg/kg.
  Arms: Dose level S8
Drug: BT-114143 — 6 subjects will receive a single dose of BT-114143 injection at 15 mg/kg.
  Arms: Dose level S9
Drug: 0.9% Sodium Chloride Injection as Placebo — Except that the S1 dose group was a pilot study group with 1 subject matched to receive a placebo, all other dose groups were each matched with 2 subjects who received placebo treatment as controls.
  Arms: control group

SUMMARY:
This study is a single-center, randomized, double-blind, placebo-controlled, single dose escalation design to evaluate the safety, tolerability, and pharmacokinetic characteristics of BT-114143 Injection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have been informed of the details of this study before the trial, have signed a written informed consent form, and voluntarily participate in the study;
* Healthy female or male subjects aged 18-55 years (inclusive) at the time of screening;
* Male subjects with a body weight of ≥50.0 kg and female subjects with a body weight of ≥45.0 kg; body mass index (BMI) ranging from 18.5 to 28 kg/m² (inclusive) [BMI = weight (kg) / height² (m²)];
* No history of abnormal eye color vision, or diseases related to the heart, liver, kidney, digestive system, nervous system, mental disorders, metabolic disorders, or blood system; those whose evaluations in terms of medical history, physical examination, vital signs, chest X-ray (posteroanterior), abdominal color Doppler ultrasound, ECG, and laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function, etc.) are normal or show mild abnormalities with no clinical significance, and are deemed eligible by the researcher.

Exclusion Criteria:

* Confirmed as COVID-19 patients or asymptomatic infected persons upon inquiry;
* Subjects who have undergone major surgery within 6 months prior to screening, or plan to undergo surgery during the study, as well as those who have previously undergone surgeries that may affect drug absorption, distribution, metabolism, or excretion (excluding appendectomy);
* Subjects with a history of or persistent arterial or venous thrombosis, or at high risk of thrombosis; those with a family history of hereditary coagulation or bleeding disorders;
* Subjects with a history of epilepsy;
* Female subjects with a history of recurrent spontaneous abortion;
* Subjects with positive hepatitis B surface antigen and/or hepatitis B e antigen, positive hepatitis C virus antibody, positive human immunodeficiency virus antibody, or positive treponema pallidum antibody;
* Subjects with a positive alcohol breath test or positive urine drug abuse screening;
* Heavy drinkers, i.e., consuming more than 14 standard units of alcohol per week within 3 months prior to screening (1 standard unit contains 14 g of alcohol, such as 360 mL of beer, 45 mL of spirits with 40% alcohol content, or 150 mL of wine);
* Subjects with a history of drug abuse (e.g., morphine, tetrahydrocannabinolic acid, methamphetamine, 3,4-methylenedioxymethamphetamine, ketamine) within 1 year prior to the trial;
* Subjects who need to take non-steroidal anti-inflammatory drugs, TXA, or blood-activating Chinese medicines (such as Panax notoginseng, Ligusticum chuanxiong, Salvia miltiorrhiza, etc.) within 1 month prior to enrollment or during the enrollment period;
* Pregnant or lactating women, or those with positive blood pregnancy test results, as well as subjects who do not agree to take effective contraceptive measures from the signing of the informed consent form until 3 months after the end of the study (see Appendix 10.1.7);
* Subjects who participated in other clinical trials and used investigational drugs within 3 months prior to the trial;
* Subjects who donated blood or lost ≥400 mL of blood within 3 months prior to the trial, or plan to donate blood or have blood components drawn during the study;
* Subjects with artificial materials in the body, such as heart valves, implants, etc., which are judged by the researcher as unsuitable for enrollment;
* Subjects with contraindications or potential risk factors for the use of TXA, including those known to be sensitive to TXA;
* Subjects who are judged by the researcher to have poor compliance, or have other factors that make them unsuitable for participating in this trial;
* Subjects who cannot complete the trial for other reasons.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2025-08-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of BT-114143 | For single administration, the follow-up will last until Day 15 after dosing; for multiple administrations, the follow-up will last until Day 21 after dosing.
  The number of Treatment-Emergent Adverse Events (TEAEs) with a severity of Grade 2 or higher in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

SECONDARY OUTCOMES:
Cmax | 15 days after administration
  Maximum Concentration
AUC | 15 days after administration
  Area Under the Concentration-Time Curve
t1/2 | 15 days after administration
  Half-Life
CL | 15 days after administration
  Clearance
Vz | 15 days after administration
  Volume of Distribution at Steady State
Changes in Plasminogen Activity Results from Baseline | 72 hours after administration
  Blood samples will be collected to determine the changes in plasminogen activation over time.
Changes in Thromboelastography (TEG) Parameters | 72 hours after administration
  Blood samples will be collect at each timepoints and TEG parameter (including R, K, Angle, MA, LY30, and CI values) will be measured to determine coagulation function of each subject.
Prothrombin Time（PT） | 15 days after administration
  the trend of change in PT from baseline
Activated Partial Thromboplastin Time（APTT） | 15 days after administration
  The change in Activated Partial Thromboplastin Time (APTT) from baseline
International Normalized Ratio（INR） | 15 days after administration
  The change in INR (International Normalized Ratio) from baseline
Fibrinogen（FIB） | 15 days after administration
  The change in FIB (Fibrinogen) from baseline
Thrombin Time（TT） | 15 days after administration
  The change in TT (Thrombin Time) from baseline
D-Dimer | 15 days after administration
  The change in D-Dimer (D-Dimer) from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- PKU Care Luzhong Hospital, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: No